CLINICAL TRIAL: NCT02110225
Title: A 24 Week Phase Ib/II, Multicenter, Randomized, Controlled, Parallel Group, Dose Ranging Study With a 24 Week Follow-up to Evaluate Safety and Potential Efficacy of 2 Doses (60, 180 µg/ml) of rhNGF Solution vs Vehicle in Patients With RP.
Brief Title: A Dose Ranging Study to Evaluate the Safety and Potential Efficacy of rhNGF in Patients With Retinitis Pigmentosa (RP)
Acronym: Lumos
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF0113; 2013-003029-26 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-12

CONDITIONS: Retinitis Pigmentosa
Keywords: Cone-Rod Degenerations; Cone-Rod Dystrophy; Cone-Rod Dystrophy 2; Cone-Rod Retinal Dystrophy; Pigmentary Retinopathy; Retinal Cone-Rod Dystrophy; Rod Cone Dystrophies; Rod-Cone Dystrophy; Tapetoretinal Degeneration
MeSH Terms: conditions — Retinitis Pigmentosa; Cone-Rod Dystrophies | interventions — cenegermin; Ophthalmic Solutions; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rhNGF 60µg/ml (Experimental): rhNGF 60 µg/ml eye drops solution, one drop 3 times a day for 24 weeks in both eyes
  Interventions: Drug: rhNGF 60 µg/ml eye drops solution
- rhNGF 180 µg/ml (Experimental): rhNGF 180 µg/ml eye drops solution, one drop 3 times a day for 24 weeks in both eyes.
  Interventions: Drug: rhNGF 180 µg/ml eye drops solution
- Vehicle (Placebo Comparator): Placebo eye drops solution, one drop 3 times a day for 24 weeks in both eyes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhNGF 60 µg/ml eye drops solution — rhNGF 60 µg/ml eye drops solution, one drop 3 times a day for 24 weeks in both eyes
  Other Names: recombinant human nerve growth factor 60 µg/ml solution
  Arms: rhNGF 60µg/ml
Drug: rhNGF 180 µg/ml eye drops solution — rhNGF 180 µg/ml eye drops solution, one drop 3 times a day for 24 weeks in both eyes
  Other Names: recombinant human nerve growth factor 180 µg/ml solution
  Arms: rhNGF 180 µg/ml
Drug: Placebo — Placebo eye drops solution, one drop 3 times a day for 24 weeks in both eyes
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of two dose regimens of recombinant human nerve growth factor (rhNGF) eye drops solution administered over 6 months versus a vehicle control in patients with typical retinitis pigmentosa. The secondary objective of this study is to attempt to show a dose response by assessing the potential efficacy of the rhNGF dose regimens for improving or slowing the deterioration of visual function outcomes at 3 and 6 months. During a 6 month follow-up period patients will be monitored to determine if there is evidence of a persistent biological effect after discontinuation of the study treatment.

DETAILED DESCRIPTION:
This is a 24-week phase Ib/II, multicenter, randomized, double-masked, vehicle controlled, parallel-group, dose-ranging study with a 24-week follow-up period to evaluate the safety and potential efficacy of two doses (60 μg/ml and 180 μg/ml) of recombinant human nerve growth factor (rhNGF) eye drops solution versus vehicle in patients with typical retinitis pigmentosa (RP).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older.
* Patients with typical forms of RP characterized by the following clinical features: classic fundus appearance (i.e. intraretinal pigment deposits, thinning and atrophy of the retinal pigment epithelium (RPE) in the mid- and far peripheral retina, with relative RPE preservation in the macula, waxy pallor of the optic disc, attenuation of the retinal vessels), reduced and delayed ERG responses, visual field constriction
* Best corrected distance visual acuity (BCDVA) score of ≥ 48 ETDRS letters (equivalent to 20/100 Snellen, +0.7 LogMar, or 0.2 decimal fraction) in either eye at the time of study enrollment.
* Documented evidence of disease progression within the 12 months prior to enrollment in the study as demonstrated by ERG (≥20% decrease in b wave amplitude in scotopic conditions or ≥25% in photopic conditions) and/or visual field testing (≥10% of Goldman Visual Field expressed as area square or ≥3 dB decrease of Humphrey Visual Field Mean Deviation).
* Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her impartial witness must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or impartial witness must have been approved by the Ethics Committee (IEC) for the current study.
* Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

* Patients with atypical, early onset (first decade) or syndromic forms of RP (e.g. paravenous, pericentral sector or unilateral RP, Leber's congenital amaurosis, Refsum disease, Usher syndrome, Bardet-Biedl syndrome, etc).
* Patients with non-recordable 30 Hz cone ERG in either eye.
* Patients with Goldman visual field less than 20º using the V4e target or residual central visual field less than -35 dB as evaluated by the 24-2 program of the Humphrey visual field in either eye.
* Evidence of an active ocular infection in either eye.
* History of uveitis or evidence of intraocular inflammation in either eye.
* History or evidence of glaucoma or an intraocular pressure (IOP) greater than or equal 21 mmHg in either eye at the time of study enrollment.
* Patients with foveal thickness ≥ 250 micrometers (as evaluated with OCT).
* History of cystoid macular oedema or presence of cystoid macular oedema on OCT at the time of study enrolment.
* Anterior segment abnormalities or media opacities obscuring the view of the posterior pole in either eye.
* History of any ocular surgery (including laser or refractive surgical procedures) in either eye within the 120 days before study enrolment. Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period.
* Treatment with corticosteroids (systemic, periocular or intravitreal) or any other non-approved, experimental, investigational or neuroprotectant therapy (systemic, topical, intravitreal) in either eye within 90 days of study enrollment.
* Use of any medication other than the study medication for the treatment of ocular diseases with the exception of artificial tears during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, PhD, Study Director — Dompé farmaceutici S.p.A., Milan
Locations (5):
- Italy (5):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera San Paolo - U.O. Oculistica, Milan
  - A.O. Seconda Università Degli Studi di Napoli - Nuovo Policlinico - UOC Oftalmologia, Naples
  - Università Cattolica del Sacro Cuore - Policlinico Gemelli - Istituto di Oftalmologia, Rome
  - IRCCS Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia, Rome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty patients were enrolled in the study. Two additional patients provided valid, written, informed consent but were not randomized due to screening failure. No study medication was administered to these patients.
Period: Overall Study
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Started | 20 | 20 | 10
Completed | 20 | 19 | 10
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle | Total
Number analyzed (Participants) | 20 | 20 | 10 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 10 | 48
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.80 (14.70) | 42.30 (10.66) | 34.90 (11.93) | 39.82 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 7 | 30
  Male | 6 | 11 | 3 | 20
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 10 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Twenty-seven patients of the Safety population experienced at least one treatment-emergent adverse event, 11 patients in the rhNGF 60 μg/ml arm, 13 patients in the rhNGF 180 μg/ml arm and 3 patients in the vehicle arm.
Time Frame: up to 48 weeks
Population: Safety population: all patients who received at least one dose of study medication. The safety population was used to analyze all safety endpoints (primary objective).
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants | 11 | 13 | 3

2. Primary Outcome: Change in Ocular Tolerability - VAS
Description: A global ocular discomfort score was determined using a 100 mm Visual Analogue Scale (VAS) on which 0 means no symptoms and 100 means the worst possible discomfort.
  Specific ocular symptoms to be assessed with the VAS included: foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, photophobia.
  For ocular tolerability analysis, mixed models for repeated measures were applied using various ocular tolerability parameters as response variable, treatment, visit and treatment by visit interaction as fixed effects, and baseline value as covariate.
Time Frame: Weeks 1, 2, 6, 12, 24
Population: Safety population: patients who received at least one dose of study medication. The safety population was used to analyze all safety endpoints (primary objective).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
units on a scale
  Foreign body sensation - Left eye, Wk 1 vs Day 0 | 5.45 (15.23) | 4.80 (21.31) | 3.50 (11.07)
  Foreign body sensation - Right eye, Wk 1 vs Day 0 | 5.75 (15.41) | 10.95 (24.44) | 4.30 (14.31)
  Foreign body sensation - Left eye, Wk 2 vs Day 0 | 3.50 (9.05) | -0.90 (13.78) | 1.10 (3.14)
  Foreign body sensation - Right eye, Wk 2 vs Day 0 | 3.55 (9.03) | 1.50 (4.89) | -0.20 (0.63)
  Foreign body sensation - Left eye, Wk 6 vs Day 0 | 4.05 (11.97) | -0.50 (9.32) | 1.70 (4.69)
  Foreign body sensation - Right eye, Wk 6 vs Day 0 | 4.05 (13.62) | 2.80 (5.91) | -0.20 (0.63)
  Foreign body sensation - Left eye, Wk 12 vs Day 0 | 2.65 (8.22) | 3.05 (15.14) | 0.60 (1.58)
  Foreign body sensation - Right eye, Wk 12 vs Day 0 | 2.45 (7.79) | 7.90 (17.13) | 0.50 (1.58)
  Foreign body sensation - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Foreign body sensation - Left eye, Wk 24 vs Day 0 | 3.35 (10.57) | 6.32 (21.14) | 1.00 (2.11)
  Foreign body sensation - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Foreign body sensation - Right eye, Wk 24 vs Day 0 | 2.94 (9.02) | 12.00 (20.11) | 0.30 (1.77)
  Burning/Stinging - Left eye, Wk 1 vs Day 0 | 4.60 (18.75) | -3.75 (18.43) | 0.20 (0.63)
  Burning/Stinging - Right eye, Wk 1 vs Day 0 | 5.85 (17.46) | 1.10 (18.39) | 0.10 (0.32)
  Burning/Stinging - Left eye, Wk 2 vs Day 0 | -0.15 (10.46) | -3.70 (20.13) | 2.20 (6.29)
  Burning/Stinging - Right eye, Wk 2 vs Day 0 | 0.25 (9.24) | -1.45 (15.15) | 2.00 (6.32)
  Burning/Stinging - Left eye, Wk 6 vs Day 0 | 4.75 (19.63) | 0.35 (16.48) | 2.80 (7.86)
  Burning/Stinging - Right eye, Wk 6 vs Day 0 | 5.60 (18.53) | 4.65 (19.59) | 2.70 (7.86)
  Burning/Stinging - Left eye, Wk 12 vs Day 0 | 6.25 (18.54) | 4.45 (21.98) | 3.30 (6.63)
  Burning/Stinging - Right eye, Wk 12 vs Day 0 | 5.30 (14.0) | 8.95 (22.77) | 3.10 (6.71)
  Burning/Stinging - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Burning/Stinging - Left eye, Wk 24 vs Day 0 | 20.35 (31.59) | 14.42 (29.15) | 1.80 (3.82)
  Burning/Stinging - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Burning/Stinging - Right eye, Wk 24 vs Day 0 | 14.82 (21.97) | 17.79 (26.13) | 1.90 (4.28)
  Itching - Left eye, Wk 1 vs Day 0 | 2.20 (17.25) | -0.95 (14.04) | 5.60 (9.20)
  Itching - Right eye, Wk 1 vs Day 0 | 2.25 (16.18) | -0.25 (12.72) | 8.90 (11.20)
  Itching - Left eye, Wk 2 vs Day 0 | -2.70 (15.59) | -1.80 (14.10) | 4.20 (6.89)
  Itching - Right eye, Wk 2 vs Day 0 | -2.50 (13.81) | -1.05 (12.59) | 2.10 (4.18)
  Itching - Left eye, Wk 6 vs Day 0 | -2.55 (15.89) | -0.25 (10.82) | 3.90 (4.43)
  Itching - Right eye, Wk 6 vs Day 0 | -2.60 (14.41) | 0.20 (8.33) | 3.10 (3.90)
  Itching - Left eye, Wk 12 vs Day 0 | -3.30 (18.94) | 3.00 (16.91) | 3.60 (7.43)
  Itching - Right eye, Wk 12 vs Day 0 | -3.70 (17.63) | 5.10 (16.45) | 2.70 (5.33)
  Itching - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Itching - Left eye, Wk 24 vs Day 0 | 2.24 (19.81) | 7.00 (19.05) | 3.00 (6.75)
  Itching - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Itching - Right eye, Wk 24 vs Day 0 | 1.53 (15.38) | 6.53 (16.41) | 2.40 (5.46)
  Ocular pain - Left eye, Wk 1 vs Day 0 | 29.95 (27.99) | 26.70 (23.91) | 0.80 (1.62)
  Ocular pain - Right eye, Wk 1 vs Day 0 | 29.50 (28.61) | 27.35 (24.63) | 0.70 (1.64)
  Ocular pain - Left eye, Wk 2 vs Day 0 | 23.45 (27.07) | 18.30 (23.20) | 2.00 (6.32)
  Ocular pain - Right eye, Wk 2 vs Day 0 | 25.50 (28.33) | 20.10 (22.58) | 2.00 (6.32)
  Ocular pain - Left eye, Wk 6 vs Day 0 | 14.10 (15.49) | 20.25 (24.56) | 0.00 (0.00)
  Ocular pain - Right eye, Wk 6 vs Day 0 | 13.90 (15.33) | 24.15 (25.83) | 0.00 (0.00)
  Ocular pain - Left eye, Wk 12 vs Day 0 | 12.60 (16.21) | 18.50 (20.00) | 3.00 (6.75)
  Ocular pain - Right eye, Wk 12 vs Day 0 | 10.40 (15.13) | 20.50 (20.24) | 5.00 (10.80)
  Ocular pain - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Ocular pain - Left eye, Wk 24 vs Day 0 | 22.94 (26.60) | 33.74 (27.72) | 1.00 (3.16)
  Ocular pain - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Ocular pain - Right eye, Wk 24 vs Day 0 | 20.12 (23.01) | 36.47 (26.07) | 1.00 (3.16)
  Sticky feeling - Left eye, Wk 1 vs Day 0 | 2.25 (23.87) | -1.40 (8.68) | 4.90 (6.51)
  Sticky feeling - Right eye, Wk 1 vs Day 0 | 2.40 (27.36) | -1.00 (8.64) | 4.50 (4.97)
  Sticky feeling - Left eye, Wk 2 vs Day 0 | -1.70 (19.76) | -2.35 (9.53) | 4.60 (6.87)
  Sticky feeling - Right eye, Wk 2 vs Day 0 | -1.15 (24.92) | -3.90 (13.47) | 4.50 (6.85)
  Sticky feeling - Left eye, Wk 6 vs Day 0 | -0.50 (19.99) | 0.75 (5.19) | 4.90 (6.92)
  Sticky feeling - Right eye, Wk 6 vs Day 0 | 0.15 (20.58) | 1.05 (6.65) | 5.10 (7.19)
  Sticky feeling - Left eye, Wk 12 vs Day 0 | -0.75 (19.49) | 2.30 (12.81) | 4.80 (6.70)
  Sticky feeling - Right eye, Wk 12 vs Day 0 | -0.15 (20.68) | 1.30 (18.11) | 5.50 (8.32)
  Sticky feeling - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Sticky feeling - Left eye, Wk 24 vs Day 0 | 3.53 (22.80) | 1.47 (13.75) | 1.00 (2.11)
  Sticky feeling - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Sticky feeling - Right eye, Wk 24 vs Day 0 | 4.12 (23.93) | 2.68 (18.44) | 1.00 (2.11)
  Blurred vision - Left eye, Wk 1 vs Day 0 | -11.45 (27.97) | -12.45 (24.46) | 1.90 (17.25)
  Blurred vision - Right eye, Wk 1 vs Day 0 | -10.50 (27.01) | -8.30 (17.09) | -0.70 (12.27)
  Blurred vision - Left eye, Wk 2 vs Day 0 | -5.70 (23.91) | -15.00 (28.27) | 1.30 (17.31)
  Blurred vision - Right eye, Wk 2 vs Day 0 | -5.35 (23.28) | -13.70 (24.75) | 1.60 (14.98)
  Blurred vision - Left eye, Wk 6 vs Day 0 | -10.50 (20.67) | -11.80 (26.36) | -1.10 (10.13)
  Blurred vision - Right eye, Wk 6 vs Day 0 | -8.95 (18.64) | -11.55 (22.53) | 0.20 (8.26)
  Blurred vision - Left eye, Wk 12 vs Day 0 | -8.20 (15.62) | -16.00 (29.26) | 0.10 (10.81)
  Blurred vision - Right eye, Wk 12 vs Day 0 | -8.40 (16.50) | -14.70 (27.66) | 0.70 (7.70)
  Blurred vision - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Blurred vision - Left eye, Wk 24 vs Day 0 | -9.35 (19.89) | -7.37 (35.28) | -1.80 (11.06)
  Blurred vision - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Blurred vision - Right eye, Wk 24 vs Day 0 | -7.82 (19.18) | -8.32 (31.21) | -1.30 (7.01)
  Photophobia - Left eye, Wk 1 vs Day 0 | -2.35 (23.33) | -6.75 (27.10) | 2.90 (18.10)
  Photophobia - Right eye, Wk 1 vs Day 0 | -1.95 (22.42) | -7.15 (27.21) | 5.10 (16.47)
  Photophobia - Left eye, Wk 2 vs Day 0 | -3.40 (17.72) | -5.90 (29.91) | -1.60 (9.02)
  Photophobia - Right eye, Wk 2 vs Day 0 | -4.05 (18.80) | -5.60 (29.66) | -0.50 (6.43)
  Photophobia - Left eye, Wk 6 vs Day 0 | -7.10 (23.16) | -8.50 (34.83) | -1.30 (10.74)
  Photophobia - Right eye, Wk 6 vs Day 0 | -6.50 (22.84) | -6.25 (36.89) | -1.70 (10.27)
  Photophobia - Left eye, Wk 12 vs Day 0 | -10.45 (22.91) | -9.80 (30.24) | -8.70 (19.86)
  Photophobia - Right eye, Wk 12 vs Day 0 | -10.60 (22.87) | -10.00 (29.69) | -7.40 (17.77)
  Photophobia - Left eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Photophobia - Left eye, Wk 24 vs Day 0 | -11.88 (29.02) | -7.37 (40.52) | -8.10 (20.01)
  Photophobia - Right eye, Wk 24 vs Day 0: number analyzed (Participants) | 17 | 19 | 10
  Photophobia - Right eye, Wk 24 vs Day 0 | -12.12 (28.23) | -8.89 (39.55) | -8.50 (19.16)

3. Primary Outcome: Change in Best Corrected Distance Visual Acuity (BCDVA) (ETDRS Chart)
Description: Best-Corrected Distance Visual Acuity (BCDVA) was assessed for each eye at each visit using an ETDRS visual acuity chart at 4 meters.
Time Frame: Weeks 1, 2, 6, 12, 24, 36, 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters read correctly
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Letters read correctly
  Week 1 vs Day 0 - left eye | 0.50 (2.86) | 1.65 (2.23) | 0.90 (2.81)
  Week 1 vs Day 0 - right eye | 1.70 (2.27) | 2.20 (3.29) | 1.70 (3.20)
  Week 2 vs Day 0 - left eye | 0.95 (2.70) | 2.15 (2.30) | 2.50 (3.10)
  Week 2 vs Day 0 - right eye | 1.40 (2.41) | 2.55 (4.24) | 2.60 (3.60)
  Week 6 vs Day 0 - left eye | 1.90 (2.73) | 1.60 (2.48) | 1.80 (3.91)
  Week 6 vs Day 0 - right eye | 1.50 (2.40) | 3.25 (4.56) | 2.00 (3.27)
  Week 12 vs Day 0 - left eye | 2.25 (3.64) | 2.50 (2.56) | 0.90 (4.46)
  Week 12 vs Day 0 - right eye | 1.85 (2.23) | 2.50 (4.47) | 1.10 (4.38)
  Week 24 vs Day 0 - left eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 vs Day 0 - left eye | 1.65 (3.90) | 2.79 (3.01) | 2.20 (3.97)
  Week 24 vs Day 0 - right eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 vs Day 0 - right eye | 2.71 (3.16) | 3.89 (5.52) | 3.60 (3.60)
  Week 36 vs Day 0 - left eye: number analyzed (Participants) | 20 | 19 | 9
  Week 36 vs Day 0 - left eye | 1.90 (4.06) | 0.47 (5.47) | 0.33 (3.28)
  Week 36 vs Day 0 - right eye: number analyzed (Participants) | 20 | 19 | 9
  Week 36 vs Day 0 - right eye | 2.15 (3.99) | 2.74 (6.62) | 0.89 (3.30)
  Week 48 vs Day 0 - left eye: number analyzed (Participants) | 20 | 19 | 10
  Week 48 vs Day 0 - left eye | 0.15 (5.32) | 0.26 (5.02) | -0.60 (3.20)
  Week 48 vs Day 0 - right eye: number analyzed (Participants) | 20 | 19 | 10
  Week 48 vs Day 0 - right eye | 1.60 (4.96) | 1.37 (6.99) | -1.00 (5.21)

4. Primary Outcome: Change in Intraocular Pressure (IOP)
Description: Intraocular Pressure was measured using either Goldmann applanation tonometry or a handheld applanation tonometer (e.g. Tonopen) after the instillation of a topical anesthetic.IOP was assessed for each eye at day 0 and at week 2, 12 and 24
Time Frame: Weeks 2,12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
mmHg
  Week 2 vs Day 0 - left eye | 0.15 (1.73) | -0.70 (2.92) | 0.30 (2.11)
  Week 2 vs Day 0 - right eye | -0.15 (1.93) | -0.40 (3.03) | 0.70 (2.11)
  Week 12 vs Day 0 - left eye | 0.55 (2.24) | -0.45 (3.35) | 0.70 (2.50)
  Week 12 vs Day 0 - right eye | 0.05 (2.06) | -0.25 (3.21) | 1.20 (2.35)
  Week 24 vs Day 0 - left eye | -0.12 (2.03) | -0.21 (2.90) | 0.00 (2.98)
  Week 24 vs Day 0 - right eye | 0.24 (2.54) | -0.53 (2.52) | 0.90 (2.13)

5. Primary Outcome: Number of Participants With Normal or Abnormal Findings by Slit Lamp Examination
Description: Slit Lamp Examination (SLE) (Biomicroscopy) was performed before the instillation of any dilating or anesthetic eye drops or fluorescein agents. SLE was executed to assess eyelids, lashes, conjunctiva, cornea, lens, iris and anterior chamber.
Time Frame: Day 0; Weeks 1, 2, 6, 12, 24, 36 and 48
Population: s
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - normal - left eye | 12 | 13 | 6
  Day 0 - abnormal - left eye | 8 | 7 | 4
  Day 0 - normal - right eye | 13 | 14 | 6
  Day 0 - abnormal - right eye | 7 | 6 | 4
  Week 1 - normal - left eye | 13 | 13 | 6
  Week 1 - abnormal - left eye | 7 | 7 | 4
  Week 1 - normal - right eye | 14 | 14 | 6
  Week 1 - abnormal - right eye | 6 | 6 | 4
  Week 2 - normal - left eye | 13 | 14 | 6
  Week 2 - abnormal - left eye | 7 | 6 | 4
  Week 2 - normal - right eye | 14 | 15 | 6
  Week 2 - abnormal - right eye | 6 | 5 | 4
  Week 6 - normal - left eye | 11 | 12 | 5
  Week 6 - abnormal - left eye | 9 | 8 | 5
  Week 6 - normal - right eye | 12 | 14 | 5
  Week 6 - abnormal - right eye | 8 | 6 | 5
  Week 12 - normal - left eye | 11 | 10 | 6
  Week 12 - abnormal - left eye | 9 | 10 | 4
  Week 12 - normal - right eye | 12 | 12 | 6
  Week 12 - abnormal - right eye | 8 | 8 | 4
  Week 24 - normal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - normal - left eye | 8 | 12 | 7
  Week 24 - abnormal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - abnormal - left eye | 9 | 7 | 3
  Week 24 - normal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - normal - right eye | 8 | 13 | 7
  Week 24 - abnormal - right eye: number analyzed (Participants) | 20 | 19 | 10
  Week 24 - abnormal - right eye | 9 | 6 | 3
  Week 36 - normal - left eye: number analyzed (Participants) | 20 | 19 | 9
  Week 36 - normal - left eye | 13 | 11 | 5
  Week 36 - abnormal - left eye: number analyzed (Participants) | 20 | 19 | 9
  Week 36 - abnormal - left eye | 7 | 8 | 4
  Week 36 - normal - right eye: number analyzed (Participants) | 20 | 19 | 9
  Week 36 - normal - right eye | 14 | 11 | 5
  Week 36 - abnormal - right eye: number analyzed (Participants) | 20 | 19 | 9
  Week 36 - abnormal - right eye | 6 | 8 | 4
  Week 48 - normal - left eye: number analyzed (Participants) | 20 | 19 | 10
  Week 48 - normal - left eye | 13 | 12 | 6
  Week 48 - abnormal - left eye: number analyzed (Participants) | 20 | 19 | 10
  Week 48 - abnormal - left eye | 7 | 7 | 4
  Week 48 - normal - right eye: number analyzed (Participants) | 20 | 19 | 10
  Week 48 - normal - right eye | 14 | 12 | 6
  Week 48 - abnormal - right eye: number analyzed (Participants) | 20 | 19 | 10
  Week 48 - abnormal - right eye | 6 | 7 | 4

6. Primary Outcome: External Ocular Examination
Description: External ocular examinations were done to assess, for each eye and at each visit, the motility of extraocular muscles, appearance and function of the eyelids.
Time Frame: Day 0, Weeks 1, 2, 6, 12, 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - normal - left eye | 20 | 19 | 9
  Day 0 - abnormal - left eye | 0 | 1 | 1
  Day 0 - normal - right eye | 20 | 19 | 10
  Day 0 - abnormal - right eye | 0 | 1 | 0
  Week 1 - normal - left eye | 20 | 19 | 10
  Week 1 - abnormal - left eye | 0 | 1 | 0
  Week 1 - normal - right eye | 20 | 19 | 10
  Week 1 - abnormal - right eye | 0 | 1 | 0
  Week 2 - normal - left eye | 20 | 19 | 10
  Week 2 - abnormal - left eye | 0 | 1 | 0
  Week 2 - normal - right eye | 20 | 19 | 10
  Week 2 - abnormal - right eye | 0 | 1 | 0
  Week 6 - normal - left eye | 19 | 19 | 10
  Week 6 - abnormal - left eye | 1 | 1 | 0
  Week 6 - normal - right eye | 20 | 19 | 10
  Week 6 - abnormal - right eye | 0 | 1 | 0
  Week 12 - normal - left eye | 20 | 19 | 10
  Week 12 - abnormal - left eye | 0 | 1 | 0
  Week 12 - normal - right eye | 20 | 18 | 10
  Week 12 - abnormal - right eye | 0 | 2 | 0
  Week 24 - normal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - normal - left eye | 17 | 18 | 10
  Week 24 - abnormal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - abnormal - left eye | 0 | 1 | 0
  Week 24 - normal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - normal - right eye | 17 | 18 | 10
  Week 24 - abnormal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - abnormal - right eye | 0 | 1 | 0

7. Primary Outcome: Change in Ocular Tolerability - Dilated Fundus Ophthalmoscopy
Description: Dilated fundus ophthalmoscopy was assessed for each eye evaluating the retina, macula, choroid and optic nerve head.
Time Frame: Day 0, Weeks 12, 24 and 48
Population: Safety population: all patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - abnormal - left eye | 20 | 20 | 10
  Day 0 - abnormal - right eye | 20 | 20 | 10
  Week 12 - abnormal - left eye | 20 | 20 | 10
  Week 12 - abnormal - right eye | 20 | 20 | 10
  Week 24 - abnormal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - abnormal - left eye | 17 | 19 | 10
  Week 24 - abnormal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Week 24 - abnormal - right eye | 17 | 19 | 10
  Week 48 - abnormal - left eye: number analyzed (Participants) | 17 | 18 | 10
  Week 48 - abnormal - left eye | 17 | 18 | 10
  Week 48 - abnormal - right eye: number analyzed (Participants) | 17 | 18 | 10
  Week 48 - abnormal - right eye | 17 | 18 | 10

8. Primary Outcome: Presence of Anti-NGF Antibodies
Description: Anti-NGF antibodies tests were performed at screening and at the end of treatment
Time Frame: At Day 0 and at week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - absent | 20 | 20 | 9
  Day 0 - missing | 0 | 0 | 1
  Week 24 - absent | 20 | 20 | 9
  Week 24 - missing | 0 | 0 | 1

9. Secondary Outcome: Change From Baseline in Contrast Sensitivity
Description: Contrast sensitivity was assessed using a Mars chart and is expressed as a log contrast sensitivity (log CS) score given by the log CS value at the lowest contrast numeral just prior to two incorrectly identified numerals, minus a scoring correction. The higher is the number of characters properly read by the patient, the higher is the contrast sensitivity.
Time Frame: Weeks 12, 24, 36 and 48
Population: Intent to treat (ITT) population: all randomized patients. The ITT population was used for the exploratory analyses of ocular parameters.
Measure: Mean (Standard Deviation); unit: score
Groups:
- rhNGF 60µg/ml: rhNGF 60 µg/ml eye drops solution, one drop 3 times a day for 24 weeks in both eyes rhNGF 60 µg/ml eye drops solution: rhNGF 60 µg/ml eye drops solution, one drop 3 times a day for 24 weeks in both eyes
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml
Number analyzed (Participants) | 20 | 20
score
  Wk 12 vs Day 0 - binocular | 0.05 (0.14) | 0.03 (0.10)
  Wk 12 vs Day 0 - left eye | 0.04 (0.17) | 0.06 (0.11)
  Wk 12 vs Day 0 - right eye | 0.03 (0.09) | 0.01 (0.17)
  Wk 24 vs Day 0 - binocular: number analyzed (Participants) | 17 | 19
  Wk 24 vs Day 0 - binocular | 0.07 (0.14) | 0.04 (0.08)
  Wk 24 vs Day 0 - left eye: number analyzed (Participants) | 17 | 19
  Wk 24 vs Day 0 - left eye | 0.09 (0.17) | 0.06 (0.13)
  Wk 24 vs Day 0 - right eye: number analyzed (Participants) | 17 | 19
  Wk 24 vs Day 0 - right eye | 0.03 (0.11) | 0.03 (0.14)
  Wk 36 vs Day 0 - binocular: number analyzed (Participants) | 20 | 19
  Wk 36 vs Day 0 - binocular | 0.05 (0.11) | -0.02 (0.11)
  Wk 36 vs Day 0 - left eye: number analyzed (Participants) | 20 | 19
  Wk 36 vs Day 0 - left eye | 0.04 (0.16) | 0.00 (0.16)
  Wk 36 vs Day 0 - right eye: number analyzed (Participants) | 20 | 19
  Wk 36 vs Day 0 - right eye | 0.06 (0.12) | -0.05 (0.18)
  Wk 48 vs Day 0 - binocular: number analyzed (Participants) | 20 | 19
  Wk 48 vs Day 0 - binocular | 0.04 (0.12) | -0.03 (0.18)
  Wk 48 vs Day 0 - left eye: number analyzed (Participants) | 20 | 19
  Wk 48 vs Day 0 - left eye | 0.08 (0.15) | -0.03 (0.21)
  Wk 48 vs Day 0 - right eye: number analyzed (Participants) | 20 | 19
  Wk 48 vs Day 0 - right eye | 0.02 (0.12) | -0.01 (0.20)

10. Secondary Outcome: Change From Baseline in Humphrey Visual Field 24-2
Description: The Humphrey Visual Field (HVF) analyzer is a tool for measuring the human visual field by providing information regarding the location of any disease processes or lesion(s) throughout the visual pathway.
  In particular, Humphrey Visual Field 24-2 was used to assess static perimetry by measuring 24 degrees temporally and 30 degrees nasally and tests 54 points.
  The Analyser projects a series of white light stimuli of varying intensities (brightness), throughout a uniformly illuminated bowl. The higher is the number of stimuli perceived by the patient, the better is the retina's ability to detect a stimulus at specific points within the visual field.
Time Frame: Weeks 12, 24, 36 and 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
dB
  Wk 12 vs Day 0 - left eye | 0.71 (2.23) | 0.48 (0.92) | 0.53 (0.68)
  Wk 12 vs Day 0 - right eye | 1.09 (2.70) | 0.80 (2.53) | 1.82 (3.20)
  Wk 24 vs Day 0 - left eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 vs Day 0 - left eye | 1.33 (4.06) | 0.20 (1.48) | -0.08 (0.75)
  Wk 24 vs Day 0 - right eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 vs Day 0 - right eye | 2.29 (3.95) | 0.13 (1.25) | 0.45 (0.95)
  Wk 36 vs Day 0 - left eye: number analyzed (Participants) | 20 | 19 | 9
  Wk 36 vs Day 0 - left eye | 1.18 (4.80) | -0.20 (0.97) | -0.13 (1.01)
  Wk 36 vs Day 0 - right eye: number analyzed (Participants) | 20 | 19 | 9
  Wk 36 vs Day 0 - right eye | 2.24 (4.73) | -0.23 (1.11) | 1.06 (2.91)
  Wk 48 vs Day 0 - left eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 vs Day 0 - left eye | 1.08 (2.61) | -0.04 (1.12) | -0.24 (1.13)
  Wk 48 vs Day 0 - right eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 vs Day 0 - right eye | 2.51 (5.29) | 0.13 (1.10) | 0.12 (2.25)

11. Secondary Outcome: Change in Goldmann Visual Field
Description: The Goldmann field exam was performed to assess kinetic perimetry on all enrolled patients.
Time Frame: Weeks 12, 24, 36 and 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
degrees
  Wk 12 vs Day 0 - left eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 12 vs Day 0 - left eye | 11.56 (27.48) | 1.27 (14.53) | 14.21 (22.92)
  Wk 12 vs Day 0 - right eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 12 vs Day 0 - right eye | 8.20 (20.37) | 3.34 (16.37) | 1.28 (25.03)
  Wk 24 vs Day 0 - left eye: number analyzed (Participants) | 16 | 18 | 10
  Wk 24 vs Day 0 - left eye | 6.47 (45.90) | 10.08 (21.02) | 15.08 (41.63)
  Wk 24 vs Day 0 - right eye: number analyzed (Participants) | 16 | 18 | 10
  Wk 24 vs Day 0 - right eye | -4.67 (35.67) | 2.00 (27.95) | 16.14 (43.97)
  Wk 36 vs Day 0 - left eye: number analyzed (Participants) | 19 | 18 | 9
  Wk 36 vs Day 0 - left eye | 2.48 (30.82) | -6.57 (28.81) | 2.37 (24.26)
  Wk 36 vs Day 0 - right eye: number analyzed (Participants) | 19 | 18 | 9
  Wk 36 vs Day 0 - right eye | -2.05 (27.77) | -11.94 (27.85) | 0.67 (25.78)
  Wk 48 vs Day 0 - left eye: number analyzed (Participants) | 19 | 18 | 10
  Wk 48 vs Day 0 - left eye | -1.79 (36.98) | -13.76 (29.37) | 6.40 (42.15)
  Wk 48 vs Day 0 - right eye: number analyzed (Participants) | 19 | 18 | 10
  Wk 48 vs Day 0 - right eye | -5.04 (28.34) | -14.49 (25.38) | 6.84 (44.01)

12. Secondary Outcome: Fundus Imaging
Description: A recordable fundus image (photo or other electronic format) showing the central 30 degrees was captured through a dilated pupil to document the appearance of the posterior pole.
Time Frame: Day 0, Weeks 24 and 48
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - normal - left eye: number analyzed (Participants) | 19 | 19 | 10
  Day 0 - normal - left eye | 1 | 0 | 0
  Day 0 - abnormal - left eye: number analyzed (Participants) | 19 | 19 | 10
  Day 0 - abnormal - left eye | 18 | 19 | 10
  Day 0 - normal - right eye: number analyzed (Participants) | 19 | 19 | 10
  Day 0 - normal - right eye | 1 | 0 | 0
  Day 0 - abnormal - right eye: number analyzed (Participants) | 19 | 19 | 10
  Day 0 - abnormal - right eye | 18 | 19 | 10
  Wk 24 - abnormal - left eye: number analyzed (Participants) | 16 | 19 | 9
  Wk 24 - abnormal - left eye | 16 | 19 | 9
  Wk 24 - abnormal - right eye: number analyzed (Participants) | 16 | 19 | 9
  Wk 24 - abnormal - right eye | 16 | 19 | 9
  Wk 48 - abnormal - left eye: number analyzed (Participants) | 17 | 18 | 10
  Wk 48 - abnormal - left eye | 17 | 18 | 10
  Wk 48 - abnormal - right eye: number analyzed (Participants) | 17 | 18 | 10
  Wk 48 - abnormal - right eye | 17 | 18 | 10

13. Secondary Outcome: Ocular Coherence Tomography (OCT)
Description: Ocular coherence tomography was performed to evaluate the cross-sectional anatomy of the macula and to document areas of retinal atrophy.
Time Frame: Day 0, Weeks 12, 24, 36 and 48
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - normal - left eye | 6 | 4 | 0
  Day 0 - abnormal - left eye | 14 | 16 | 10
  Day 0 - normal - right eye | 7 | 4 | 0
  Day 0 - abnormal - right eye | 13 | 16 | 10
  Wk 12 - normal - left eye | 7 | 2 | 0
  Wk 12 - abnormal - left eye | 13 | 18 | 10
  Wk 12 - normal - right eye | 8 | 3 | 0
  Wk 12 - abnormal - right eye | 12 | 17 | 10
  Wk 24 - normal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 - normal - left eye | 2 | 1 | 2
  Wk 24 - abnormal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 - abnormal - left eye | 15 | 18 | 8
  Wk 24 - normal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 - normal - right eye | 3 | 2 | 2
  Wk 24 - abnormal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 - abnormal - right eye | 14 | 17 | 8
  Wk 36 - normal - left eye: number analyzed (Participants) | 18 | 19 | 9
  Wk 36 - normal - left eye | 4 | 3 | 0
  Wk 36 - abnormal - left eye: number analyzed (Participants) | 18 | 19 | 9
  Wk 36 - abnormal - left eye | 14 | 16 | 9
  Wk 36 - normal - right eye: number analyzed (Participants) | 18 | 19 | 9
  Wk 36 - normal - right eye | 5 | 3 | 0
  Wk 36 - abnormal - right eye: number analyzed (Participants) | 18 | 19 | 9
  Wk 36 - abnormal - right eye | 13 | 16 | 9
  Wk 48 - normal - left eye: number analyzed (Participants) | 19 | 19 | 10
  Wk 48 - normal - left eye | 2 | 3 | 0
  Wk 48 - abnormal - left eye: number analyzed (Participants) | 19 | 19 | 10
  Wk 48 - abnormal - left eye | 17 | 16 | 10
  Wk 48 - normal - right eye: number analyzed (Participants) | 19 | 19 | 10
  Wk 48 - normal - right eye | 2 | 3 | 0
  Wk 48 - abnormal - right eye: number analyzed (Participants) | 19 | 19 | 10
  Wk 48 - abnormal - right eye | 17 | 16 | 10

14. Secondary Outcome: Microperimetry
Description: MP1 microperimetry was analyzed to provide a more accurate measurement of retinal sensitivity in the central visual field, even in patients with unstable or extrafoveal fixation.
Time Frame: Day 0, Weeks 12, 24, 36 and 48
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - normal - left eye: number analyzed (Participants) | 18 | 19 | 10
  Day 0 - normal - left eye | 1 | 1 | 1
  Day 0 - abnormal - left eye: number analyzed (Participants) | 18 | 19 | 10
  Day 0 - abnormal - left eye | 17 | 18 | 9
  Day 0 - normal - right eye: number analyzed (Participants) | 18 | 19 | 10
  Day 0 - normal - right eye | 2 | 2 | 1
  Day 0 - abnormal - right eye: number analyzed (Participants) | 18 | 19 | 10
  Day 0 - abnormal - right eye | 16 | 17 | 9
  Week 12 - normal - left eye: number analyzed (Participants) | 15 | 14 | 8
  Week 12 - normal - left eye | 0 | 1 | 1
  Week 12 - abnormal - left eye: number analyzed (Participants) | 15 | 14 | 8
  Week 12 - abnormal - left eye | 15 | 13 | 7
  Week 12 - normal - right eye: number analyzed (Participants) | 15 | 14 | 8
  Week 12 - normal - right eye | 2 | 1 | 1
  Week 12 - abnormal - right eye: number analyzed (Participants) | 15 | 14 | 8
  Week 12 - abnormal - right eye | 13 | 13 | 7
  Week 24 - normal - left eye: number analyzed (Participants) | 14 | 18 | 9
  Week 24 - normal - left eye | 0 | 1 | 1
  Wk 24 - abnormal - left eye: number analyzed (Participants) | 14 | 18 | 9
  Wk 24 - abnormal - left eye | 14 | 17 | 8
  Wk 24 - normal - right eye: number analyzed (Participants) | 14 | 18 | 9
  Wk 24 - normal - right eye | 1 | 2 | 1
  Wk 24 - abnormal - right eye: number analyzed (Participants) | 14 | 18 | 9
  Wk 24 - abnormal - right eye | 13 | 16 | 8
  Wk 36 - normal - left eye: number analyzed (Participants) | 19 | 17 | 9
  Wk 36 - normal - left eye | 0 | 2 | 1
  Wk 36 - abnormal - left eye: number analyzed (Participants) | 19 | 17 | 9
  Wk 36 - abnormal - left eye | 19 | 15 | 8
  Wk 36 - normal - right eye: number analyzed (Participants) | 19 | 17 | 9
  Wk 36 - normal - right eye | 0 | 1 | 0
  Week 36 - abnormal - right eye: number analyzed (Participants) | 19 | 17 | 9
  Week 36 - abnormal - right eye | 19 | 16 | 9
  Wk 48 - normal - left eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 - normal - left eye | 1 | 1 | 1
  Wk 48 - abnormal - left eyew: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 - abnormal - left eyew | 19 | 18 | 9
  Wk 48 - normal - right eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 - normal - right eye | 1 | 1 | 1
  Wk 48 - abnormal - right eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 - abnormal - right eye | 19 | 18 | 9

15. Secondary Outcome: Binocular Estermann Visual Field
Description: Binocular visual field with Estermann grid testing a stimulus array of 120 points spread over an area extending approximately ±75° horizontally, 35° superiorly and 55° inferiorly while the patient looked steadily at the fixation target.
Time Frame: Day 0, Weeks 12, 24, 36 and 48
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - normal: number analyzed (Participants) | 19 | 20 | 10
  Day 0 - normal | 1 | 2 | 2
  Day 0 - abnormal: number analyzed (Participants) | 19 | 20 | 10
  Day 0 - abnormal | 18 | 18 | 8
  Wk 12 - normal: number analyzed (Participants) | 18 | 19 | 10
  Wk 12 - normal | 0 | 2 | 1
  Wk 12 - abnormal: number analyzed (Participants) | 18 | 19 | 10
  Wk 12 - abnormal | 18 | 17 | 9
  Wk 24 - abnormal: number analyzed (Participants) | 15 | 17 | 8
  Wk 24 - abnormal | 15 | 17 | 8
  Wk 36 - abnormal: number analyzed (Participants) | 16 | 15 | 8
  Wk 36 - abnormal | 16 | 15 | 8
  Wk 48 - normal: number analyzed (Participants) | 19 | 19 | 10
  Wk 48 - normal | 1 | 0 | 1
  Wk 48 - abnormal: number analyzed (Participants) | 19 | 19 | 10
  Wk 48 - abnormal | 18 | 19 | 9

16. Secondary Outcome: Electrorethinogram (ERG)
Description: A full field and 30 Hz flicker ERG was performed according to international standards. Patients were treated with anesthetic and dilating drops prior to the ERG procedure.
Time Frame: Day 0, Weeks 12, 24, 36 and 48
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Day 0 - abnormal - left eye | 20 | 20 | 10
  Day 0 - abnormal - right eye | 20 | 20 | 10
  Wk 12 - abnormal - left eye: number analyzed (Participants) | 18 | 20 | 10
  Wk 12 - abnormal - left eye | 18 | 20 | 10
  Wk 12 - abnormal - right eye: number analyzed (Participants) | 18 | 20 | 10
  Wk 12 - abnormal - right eye | 18 | 20 | 10
  Wk 24 - abnormal - left eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 - abnormal - left eye | 17 | 19 | 10
  Wk 24 - abnormal - right eye: number analyzed (Participants) | 17 | 19 | 10
  Wk 24 - abnormal - right eye | 17 | 19 | 10
  Wk 36 - abnormal - left eye: number analyzed (Participants) | 18 | 19 | 9
  Wk 36 - abnormal - left eye | 18 | 19 | 9
  Wk 36 - abnormal - right eye: number analyzed (Participants) | 18 | 19 | 9
  Wk 36 - abnormal - right eye | 18 | 19 | 9
  Wk 48 - abnormal - left eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 - abnormal - left eye | 20 | 19 | 10
  Wk 48 - abnormal - right eye: number analyzed (Participants) | 20 | 19 | 10
  Wk 48 - abnormal - right eye | 20 | 19 | 10

ADVERSE EVENTS:
Time Frame: Weeks 1, 2, 6, 12 and 24, plus follow-up at weeks 36 and 48
Arm/Group | rhNGF 60µg/ml | rhNGF 180 µg/ml | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 11/20 | 13/20 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 60µg/ml (N=20) | rhNGF 180 µg/ml (N=20) | Vehicle (N=10)
ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rhNGF 60µg/ml (N=20) | rhNGF 180 µg/ml (N=20) | Vehicle (N=10)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Corneal epitelium defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 4 (4) | 0 (0)
Eye pain (Eye disorders) | 6 (6) | 8 (8) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Night blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
LImitations and caveats non specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No